CLINICAL TRIAL: NCT03755414
Title: A Single-Arm, Open-Label, Pilot Study and Expansion Study of JAK Inhibitor Itacitinib for the Prophylaxis of Graft-Versus-Host Disease and Cytokine Release Syndrome After T-cell Replete Haploidentical Peripheral Blood Hematopoietic Cell Transplantation
Brief Title: Study of Itacitinib for the Prophylaxis of Graft-Versus-Host Disease and Cytokine Release Syndrome After T-cell Replete Haploidentical Peripheral Blood Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Incyte Corporation (Industry); American Society of Hematology (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201903114; K12CA167540 (NIH)
Record Dates: First submitted 2018-11-20; First posted 2018-11-28 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndromes; Non-Hodgkin Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Stem Cell Transplantation; itacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Pilot Study: Itacitinib (Experimental): * Will undergo institutionally standard myeloablative or reduced intensity chemotherapy or chemoradiotherapy
  * Stem cell transplantation on Day 0
  * Itacitinib 200 mg/day from Day -3 to Day 100. After Day 100, for patients at a dose of 200 mg daily, reduce to 100 mg daily for 1 month, then every other day for one month, then discontinue OR after day 100, for patients already dose reduced to 100 mg daily, reduce to 100 mg every other day then discontinue OR after day 100, for patients on study drug hold, discontinue permanently
  * To address concerns of engraftment failure using itacitinib throughout the transplant period, for the first three patients the investigators will consent the donor for a second CD34+ collection to use as a rescue in the case of engraftment failure.
  Interventions: Procedure: Stem cell transplantation; Drug: Itacitinib; Other: Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT); Other: Human Activity Profile
- Expansion Phase: Itacitinib (Experimental): * Will undergo institutionally standard myeloablative or reduced intensity chemotherapy or chemoradiotherapy
  * Stem cell transplantation on Day 0
  * Itacitinib 200 mg/day from Day -3 to Day 180. After Day 180, for patients at a dose of 200 mg daily, reduce to 100 mg daily for 1 month, then every other day for one month, then discontinue OR after day 180, for patients already dose reduced to 100 mg daily, reduce to 100 mg every other day then discontinue OR after day 180, for patients on study drug hold, discontinue permanently
  Interventions: Procedure: Stem cell transplantation; Drug: Itacitinib; Other: Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT); Other: Human Activity Profile
- Donors (No Intervention): -Donors were consented for the patients enrolled in the Safety Lead-In Phase (planned 3 patients). Donors were consented for a second CD34+ collection to use as a rescue in the case of engraftment failure and for collection of a research blood specimen prior to mobilization.

INTERVENTIONS:
Procedure: Stem cell transplantation — Standard of care
  Arms: Expansion Phase: Itacitinib; Pilot Study: Itacitinib
Drug: Itacitinib — Itacitinib may be taken without regard to food.
  Arms: Expansion Phase: Itacitinib; Pilot Study: Itacitinib
Other: Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) — * Screening, day 14, day 28, day 42, day 74, day 100, taper period, and follow-up (pilot study)
  * Screening, day 14, day 28, day 42, day 74, day 100, day 180, taper period, and follow-up period (expansion study)
  Arms: Expansion Phase: Itacitinib; Pilot Study: Itacitinib
Other: Human Activity Profile — * Screening, day 14, day 28, day 42, day 74, day 100, taper period, and follow-up (pilot study)
  * Screening, day 14, day 28, day 42, day 60, day 74, day 100, day 180, taper period, and follow-up period (expansion study)
  Arms: Expansion Phase: Itacitinib; Pilot Study: Itacitinib

SUMMARY:
In this trial, the investigators will begin to explore the possibility that, as in mice, janus kinase inhibitor 1 (JAK1) inhibition with haploidentical-hematopoietic cell transplantation (HCT) may mitigate graft-versus-host-disease (GVHD) and cytokine release syndrome (CRS) while retaining Graft-versus-Leukemia (GVL) and improving engraftment. The purpose of this pilot study is to determine the safety of itacitinib with haplo-hematopoietic cell transplantation (HCT) measured by the effect on engraftment and grade III-IV GVHD.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria within 30 days prior to Day 0 unless otherwise noted.

* Diagnosis of a hematological malignancy listed below:

  * Acute myelogenous leukemia (AML) in complete morphological remission (based on International Working Group (IWG) Criteria)
  * Acute lymphocytic leukemia (ALL) in complete morphological remission (MRD negative, based on IWG Criteria)
  * Myelodysplastic syndrome with ≤ 5% blasts in bone marrow.
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete or partial remission.
* Planned treatment is myeloablative or reduced intensity conditioning followed by T Cell-replete peripheral blood haploidentical donor transplantation
* Available human leukocyte antigen (HLA)-haploidentical donor who meets the following criteria:

  * Blood-related family member, including (but not limited to) sibling, offspring, cousin, nephew, or parent. Younger donors should be prioritized.
  * At least 18 years of age
  * HLA-haploidentical donor/recipient match by at least low-resolution typing per institutional standards.
  * In the investigator's opinion, is in general good health, and medically able to tolerate leukapheresis required for harvesting hematopoietic stem cells (HSC).
  * No active hepatitis.
  * Negative for human T-cell lymphotrophic virus (HTLV) and human immunodeficiency virus (HIV).
  * Not pregnant.
  * Safety Lead-In Phase: For the first three patients, the donor must consent to a second product collection should it prove necessary.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ function as defined below:

  * Total bilirubin must be within normal range at baseline
  * Aspartate aminotransferase (AST)(SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 3.0 x institutional upper limit of normal (IULN).
  * Creatinine ≤ 1.5 x IULN OR creatinine clearance ≥ 45 mL/min/1.73 m^2 by Cockcroft-Gault Formula.
  * Oxygen saturation ≥ 90% on room air.
  * Left ventricular ejection fraction (LVEF) ≥ 40%.
  * Forced expiratory volume (FEV1) and forced vital capacity (FVC) ≥ 40% predicted, diffusing capacity of the lung for carbon monoxide (DLCOc) ≥ 40% predicted. If DLCO is < 40%, patients will still be considered eligible if deemed safe after a pulmonary evaluation.
* At least 18 years of age at the time of study registration
* Able to understand and willing to sign an Institutional Review Board (IRB) approved written informed consent document (or that of legally authorized representative, if applicable).
* Must be able to receive GVHD prophylaxis with tacrolimus, mycophenolate mofetil, and cyclophosphamide

Exclusion Criteria:

* Must not have undergone a prior allogeneic donor (related, unrelated, or cord) transplant. Prior autologous transplant is not exclusionary.
* Presence of donor-specific antibodies (DSA) with Mean Fluorescence Intensity (MFI) of ≥2000 as assessed by the single antigen bead assay.
* Known HIV or active hepatitis B or C infection.
* Known hypersensitivity to one or more of the study agents, including Ruxolitinib and Itacitinib.
* Must not have myelofibrosis (unless they are enrolled Amendment #5 or later) or other disease known to prolong neutrophil engraftment to > 35 days after transplant.
* Must not receive antithymocyte globulin as part of pre-transplant conditioning regimens.
* Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug (Day -3).
* Pregnant and/or breastfeeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disease, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
* Immunosuppressive doses of steroids. Subjects with steroids for adrenal insufficiency will not be excluded.

Additional Inclusion Criteria Under Amendment 5

* Five subjects with myelofibrosis will be enrolled in the expansion phase.
* Three patients whose donors fail to collect the target number of CD34+ cells and the treating physician choses to move forward with the haplo-HCT will be enrolled in the expansion phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Abboud, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The study protocol will also be made available. Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary"), for the purpose of achieving their approved aims. Patient who opt out of data sharing will not be included.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 9 months and ending 36 months following article publication

REFERENCES:
- [Derived] Abboud R, Schroeder MA, Rettig MP, Jayasinghe RG, Gao F, Eisele J, Gehrs L, Ritchey J, Choi J, Abboud CN, Pusic I, Jacoby M, Westervelt P, Christopher M, Cashen A, Ghobadi A, Stockerl-Goldstein K, Uy GL, DiPersio JF. Itacitinib for prevention of graft-versus-host disease and cytokine release syndrome in haploidentical transplantation. Blood. 2025 Mar 27;145(13):1382-1394. doi: 10.1182/blood.2024026497. PMID 39576962
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
Started | 22 | 27 | 6
Completed | 20 | 25 | 4
Not Completed | 2 | 2 | 2
Not completed — Did not continue with treatment due to low donor collection | 2 | 1 | 0
Not completed — Recipient did not continue with treatment due to low donor cell collection | 0 | 0 | 2
Not completed — Non-compliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors | Total
Number analyzed (Participants) | 22 | 27 | 6 | 55
Age, Continuous [Median (Full Range); unit: years] | 57.5 [20 to 73] | 61 [19 to 72] | 37.5 [27 to 45] | 58 [19 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 2 | 21
  Male | 12 | 18 | 4 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 21 | 27 | 6 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 2 | 0 | 4
  White | 18 | 25 | 6 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 27 | 6 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Graft Failure (Pilot Study Only)
Description: Failure to engraft will be defined as failure to achieve absolute neutrophil count >500 for 3 days by day 35.
Time Frame: By day 35
Population: Donors and participants in the Expansion Phase were not evaluable for this outcome measure. There were 2 participants in the Pilot Study who were not evaluable due to not continuing with treatment due to low donor collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
Number analyzed (Participants) | 20 | 0 | 0
Participants | 0 |  |

2. Primary Outcome: Number of Participants With Grades III-IV Acute GVHD
Description: -Incidence of acute grade III-IV GVHD will be assessed using Mount Sinai Acute GvHD International Consortium (MAGIC) criteria. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Time Frame: Through day 100
Population: Donors were not evaluable for this outcome measure. There were 2 participants in the Pilot Study and 2 participants in the Expansion Phase who were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
Number analyzed (Participants) | 20 | 25 | 0
Participants | 0 | 0 |

3. Secondary Outcome: Number of Participants Who Experience Cytokine Release Syndrome (CRS)
Description: * The number of participants who experience CRS will be summarized by count of participants who experience Grade 1, 2, 3, 4, & 5 CRS. The worst grade experienced by participant will be noted.
  * Grade 1: symptoms not life threatening & require symptomatic treatment alone, includes fever, nausea, fatigue, malaise
  * Grade 2: symptoms require/respond to limited intervention - oxygen (O2) <40%, <=3 liters (L) nasal cannula or hypotension responsive to fluids or low dose of 1 vasopressor or grade 2 renal or hepatic toxicity
  * Grade 3: symptoms require/respond to aggressive intervention - O2 >=40%, >3L nasal cannula or hypotension requiring high dose or multiple vasopressors or grade 3 renal toxicity or grade 4 transaminitis, new onset altered mental status, new cardiomyopathy without wall motion abnormality
  * Grade 4: life-threatening symptoms - requirement for ventilator support or grade 4 rental toxicity (excluding transaminitis)
  * Grade 5: death
Time Frame: Through day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
Number analyzed (Participants) | 20 | 25 | 0
Participants
  Grade 1 or above | 18 | 15 |
  Grade 2 or above | 5 | 1 |

4. Secondary Outcome: Number of Participants With Treatment Related Mortality
Description: -Death that results from a transplant procedure-related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause
Time Frame: Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
Number analyzed (Participants) | 20 | 25 | 0
Participants | 0 | 0 |

5. Secondary Outcome: Cumulative Incidence of Grades II-IV Acute GVHD (Expansion Phase)
Description: * Incidence of acute grade II-IV GVHD will be assessed using Mount Sinai Acute GvHD International Consortium (MAGIC) criteria. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
  * The cumulative incidence of aGVHD was estimated using Fine-Gray's sub-distribution methods to account for competing risk of death without aGVHD.
Time Frame: Day 100
Population: Donors and participants in the Pilot Phase are not evaluable for this outcome measure. There were 2 participants in the Expansion Phase who were not evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
Number analyzed (Participants) | 0 | 25 | 0
percent |  | 20 [7 to 38] |

ADVERSE EVENTS:
Time Frame: - Adverse events (AEs) were tracked from start of itacitinib through 30 days after last dose (median length of follow-up 166 days, full range 16-287 days). - All-cause mortality was collected from start of itacitinib through completion of follow-up (up to day 365).
Description: * SAEs, AEs and all-cause mortality were not collected on donors.
  * The protocol contains the selected AEs that were collected for those in the pilot and expansion phase.
  * SAEs and AEs were collected on any patient who received at least one dose of itacitinib.
  * All-cause morality was collected for any patient who completed were compliant with the assigned treatment.
Arm/Group | Pilot Study: Itacitinib | Expansion Phase: Itacitinib | Donors
All-Cause Mortality (participants affected / at risk) | 3/20 | 8/25 | 0/0
Serious Adverse Events (participants affected / at risk) | 14/20 | 24/26 | 0/0
Other Adverse Events (participants affected / at risk) | 20/20 | 26/26 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot Study: Itacitinib (N=20) | Expansion Phase: Itacitinib (N=26) | Donors (N=0)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | NA
Diarrhea (Gastrointestinal disorders) | 3 | 0 | NA
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | NA
Nausea (Gastrointestinal disorders) | 2 | 2 | NA
Fever (General disorders) | 1 | 4 | NA
Adenovirus (Infections and infestations) | 1 | 0 | NA
CMV viremia (Infections and infestations) | 1 | 0 | NA
COVID-19 infection (Infections and infestations) | 0 | 1 | NA
Enterococcus bacteremia (Infections and infestations) | 0 | 1 | NA
Enterocolitis infectious (Infections and infestations) | 2 | 3 | NA
HSV stomatitis (Infections and infestations) | 1 | 0 | NA
Lung infection (Infections and infestations) | 4 | 5 | NA
MSSA bacteremia septic arthritis (Infections and infestations) | 0 | 1 | NA
RSV infection (Infections and infestations) | 0 | 1 | NA
Sepsis (Infections and infestations) | 1 | 2 | NA
Skin infection (Infections and infestations) | 0 | 2 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Relapsed disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | NA
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | NA
Cystitis noninfective (Renal and urinary disorders) | 1 | 1 | NA
Hematuria (Renal and urinary disorders) | 1 | 0 | NA
Renal colic (Renal and urinary disorders) | 1 | 0 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot Study: Itacitinib (N=20) | Expansion Phase: Itacitinib (N=26) | Donors (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 13 | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | NA
Colitis (Gastrointestinal disorders) | 1 | 0 | NA
Dysphagia (Gastrointestinal disorders) | 0 | 1 | NA
Esophagitis (Gastrointestinal disorders) | 0 | 1 | NA
Mucositis oral (Gastrointestinal disorders) | 7 | 5 | NA
Nausea (Gastrointestinal disorders) | 0 | 1 | NA
Rectal pain (Gastrointestinal disorders) | 0 | 1 | NA
Cytokine release syndrome (Immune system disorders) | 1 | 0 | NA
BK virus (Infections and infestations) | 1 | 0 | NA
Enterococcus faecium bacteremia (Infections and infestations) | 0 | 1 | NA
Enterocolitis infectious (Infections and infestations) | 0 | 1 | NA
Lung infection (Infections and infestations) | 1 | 1 | NA
Paronychia (Infections and infestations) | 1 | 0 | NA
Sepsis (Infections and infestations) | 1 | 2 | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | NA
Alanine aminotransferase increased (Investigations) | 2 | 4 | NA
Alkaline phosphatase increased (Investigations) | 0 | 2 | NA
Aspartate aminotransferase increased (Investigations) | 1 | 3 | NA
Creatinine increased (Investigations) | 0 | 1 | NA
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 2 | NA
Lymphocyte count decreased (Investigations) | 2 | 13 | NA
Neutrophil count decreased (Investigations) | 19 | 18 | NA
Platelet count decreased (Investigations) | 19 | 16 | NA
Weight loss (Investigations) | 0 | 2 | NA
White blood cell decreased (Investigations) | 20 | 17 | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 5 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA
Encephalopathy (Nervous system disorders) | 0 | 1 | NA
Headache (Nervous system disorders) | 1 | 1 | NA
Tremor (Nervous system disorders) | 1 | 0 | NA
Insomnia (Psychiatric disorders) | 0 | 3 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | NA
Renal calculi (Renal and urinary disorders) | 1 | 0 | NA
Hypotension (Vascular disorders) | 0 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03755414/Prot_SAP_001.pdf
  • Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03755414/ICF_002.pdf